CLINICAL TRIAL: NCT02758210
Title: Evaluating the Electro Magnetic Interference of Using Tablet and Smart Phone on Leadless Pacemaker (MICRA)
Acronym: MICRA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Mikhael El Chami, Associate Professor, Emory University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: IRB00084576
Record Dates: First submitted 2016-04-19; First posted 2016-05-02 (Estimated); Results first posted 2017-10-02 (Actual); Last update posted 2017-11-09 (Actual); Status verified 2017-10

CONDITIONS: Bradycardia, Atrial Tachyarrhythmia
Keywords: Bradycardia; Atrial Tachyarrhythmia; Smart Phone; Tablet
MeSH Terms: conditions — Bradycardia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Participants with MICRA Device (Experimental): Participants that received the MICRA device prior to study enrollment will have monitored use of Smart Phone and Tablet at one study visit. Electrogram printing will take place during use of each device to see if there is any pacing inhibition or asynchronous pacing.
  Interventions: Device: Use of a Tablet; Device: Use of a Smart Phone

INTERVENTIONS:
Device: Use of a Tablet — Testing of the electromagnetic field exposure and it's affect on the participant's previously implanted MICRA device is assessed by interrogation of the device before using Tablet and while using the Tablet. The measured position of the Tablets tested will be normal routine position (noting at least 6 inches/15 centimeters from their pacemaker).
Device: Use of a Smart Phone — Testing of the electromagnetic field exposure and it's affect on the participant's previously implanted MICRA device is assessed by interrogation of the device before using a Smart phone and while using the Smart phone. The position of the Smart phone tested will be normal position at the ear and while texting (noting at least 6 inches/15 centimeters from their pacemaker).

SUMMARY:
The purpose of this study is to evaluate the effects that electromagnetic field exposure from using a tablet and smart phone have on a leadless pacemaker (MICRA device).

DETAILED DESCRIPTION:
With advancement in technology, people are exposed to new sources of electromagnetic field like tablets and smart phones. There are magnets in smart phones and tablets that could affect the functions of pacemakers. The main purpose of this study is to evaluate the effects of electromagnetic field exposure from using a tablet and a smart phone with participants that have a leadless pacemaker (MICRA device) implanted inside them. Participants will be asked to report any symptoms that they experience during the testing.

ELIGIBILITY:
Inclusion Criteria:

* Patients enrolled in MICRA Study and MICRA CA study at Emory University Hospital and Emory Midtown Hospital
* Able to consent

Exclusion Criteria:

* Patients not enrolled in MICRA Study and MICRA CA study at Emory University Hospital and Emory Midtown Hospital
* Children and vulnerable populations

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2016-04; Primary Completion 2016-10-24 (Actual); Study Completion 2016-10-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mikhael El Chami, MD, Principal Investigator — Emory University
Locations (2):
- United States (2):
  - Emory University Hospital Midtown, Atlanta, Georgia
  - Emory University Hospital, Atlanta, Georgia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from those already participating in the MICRA Study and MICRA CA Study at Emory University Hospital and Emory University Hospital Midtown. Participants for this substudy were enrolled between April 2016 and October 2016.
Groups:
- Participants With MICRA Device: Participants that received the MICRA device prior to study enrollment and who consented to having monitored use of a smart phone and a tablet at a single study visit.
Period: Overall Study
Arm/Group | Participants With MICRA Device
Started | 20
Completed | 20
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Patients who were eligible to participate and were randomized to a study arm
Arm/Group | Participants With MICRA Device
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 19
Age, Continuous [Mean (Standard Deviation); unit: years] | 78.9 (9.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 20
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 9
  White | 11
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 20
Hypertension [Count of Participants; unit: Participants] — Participants with a diagnosis of hypertension
  Participants | 17
Diabetes [Count of Participants; unit: Participants] — Participants with a diagnosis of diabetes
  Participants | 8
Congestive heart failure [Count of Participants; unit: Participants] — Participants with a diagnosis of congestive heart failure
  Participants | 6
Pacing indication: permanent atrial fibrillation and high-grade AV block [Count of Participants; unit: Participants] | 10
Atrioventricular (AV) node ablation concomitantly with the MICRA procedure [Count of Participants; unit: Participants] | 5

OUTCOME MEASURES:

1. Primary Outcome: Device Response Assessed by Asynchronous Pacing When Using a Smart Phone
Description: Cardiac pacing before and during use of a smart phone was monitored to assess asynchronous pacing due to electromagnetic field exposure. The initial programmed pacing settings of the MICRA device are compared to any changes during the smart phone usage.
Time Frame: Baseline (Before use of Smart Phone), During use of Smart Phone (an average of 5 minutes)
Measure: Mean (Standard Deviation); unit: ohms
Arm/Group | Participants With MICRA Device
Number analyzed (Participants) | 20
ohms
  Before Smart Phone Use | 528 (88)
  During Smart Phone Use | 547 (87)

2. Primary Outcome: Number of Participants Experiencing Asynchronous Pacing While Using a Tablet
Description: Cardiac pacing before and during use of a tablet were monitored to assess if there is asynchronous pacing due to electromagnetic field exposure. The initial programmed pacing settings of the MICRA device are compared to any changes during the tablet usage.
Time Frame: Baseline (Before use of Tablet), During use of Tablet (an average of 5 minutes)
Measure: Count of Participants; unit: Participants
Arm/Group | Participants With MICRA Device
Number analyzed (Participants) | 20
Participants
  Asynchronous Pacing Before Tablet Use | 0
  Asynchronous Pacing During Tablet Use | 0

3. Primary Outcome: Number of Participants Experiencing Inhibition of Ventricular Pacing While Using a Smart Phone
Description: Ventricular pacing before and during use of a smart phone was monitored to assess the presence of inhibition of ventricular pacing due to electromagnetic field exposure. The programmed pacing of the MICRA device is specific for each participant. The individualized, initial programmed pacing settings of the MICRA device are compared to any changes during the smart phone usage.
Time Frame: Baseline (Before use of Smart Phone), During use of Smart Phone (an average of 5 minutes)
Measure: Count of Participants; unit: Participants
Arm/Group | Participants With MICRA Device
Number analyzed (Participants) | 20
Participants | 0

4. Primary Outcome: Device Response While Using a Tablet, Assessed by Ventricular Pacing
Description: Ventricular pacing before and during use of a tablet was monitored to assess if there's inhibition of ventricular pacing due to electromagnetic field exposure. The initial programmed pacing settings of the MICRA device are compared to any changes during the tablet usage. The assessment of this outcome measure takes an average of 5 minutes.
Time Frame: Baseline (Before use of Tablet), During use of Tablet (an average of 5 minutes)
Measure: Mean (Standard Deviation); unit: millivolts (mV)
Arm/Group | Participants With MICRA Device
Number analyzed (Participants) | 20
millivolts (mV)
  Sensing Amplitude Before Tablet Use | 10.8 (4.7)
  Sensing Amplitude During Tablet Use | 11 (4.8)

5. Secondary Outcome: Number of Participants Reporting Clinical Symptoms While Using a Smart Phone
Description: Participants were asked to report any clinical symptoms that they experienced when using the smart phone.
Time Frame: Baseline (Before use of Smart Phone), During use of Smart Phone (an average of 5 minutes)
Measure: Count of Participants; unit: Participants
Arm/Group | Participants With MICRA Device
Number analyzed (Participants) | 20
Participants | 0

6. Secondary Outcome: Number of Participants Reporting Clinical Symptoms While Using a Tablet
Description: Participants were asked to report any clinical symptoms that they experienced when using the tablet.
Time Frame: Baseline (Before use of Tablet), During use of Tablet (an average of 5 minutes)
Measure: Count of Participants; unit: Participants
Arm/Group | Participants With MICRA Device
Number analyzed (Participants) | 20
Participants | 0

ADVERSE EVENTS:
Time Frame: Participants reported any adverse events from the time of consenting to take part in the study throughout the duration of the study activities. All study activities were performed in a single study visit.
Arm/Group | Participants With MICRA Device
All-Cause Mortality (participants affected / at risk) | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes